CLINICAL TRIAL: NCT04372264
Title: Comparison of the Effect of Intravenous Paracetamol, Dexketoprofen and Ibuprofen on Visual Analogue Scale (VAS) in the Treatment of Acute Migraine Attack Headache in the Emergency Department: A Double-Blinded, Randomized, Controlled Trial
Brief Title: Intravenous Paracetamol, Dexketoprofen and Ibuprofen in the Treatment of Acute Migraine Attack Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ibrahim Turkcuer, Professor, MD, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019TIPF006
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-05

CONDITIONS: Headache, Migraine
Keywords: paracetamol; dexketoprofen; ibuprofen; emergency department; migraine attack headache
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Acetaminophen; dexketoprofen trometamol; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracetamol (Experimental): 1000 mg of paracetamol ( perfalgan 10mg/ml solutionBristol- Myers Squibb_UK) intravenous (IV) was given 70 patients,
  Interventions: Drug: Paracetamol
- Dexketoprofen (Experimental): Second Group: dexketoprofen 50 mg ( arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 70 patients,
  Interventions: Drug: Dexketoprofen
- Ibuprofen (Experimental): third group: 400 mg Ibuprofen (İntrafen 400 mg vial-Gen-İstanbul) intravenous (IV) was given 70 patients, which determined to be applied as a group.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg of paracetamol ( perfalgan 10mg/ml solutionBristol- Myers Squibb_UK) intravenous (IV) was given 70 patients,
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Dexketoprofen — Second Group: dexketoprofen 50 mg ( arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 70 patients,
  Other Names: ASEKET; DARKIN; DEXALGIN; DESTIYO; DEXCORIL
  Arms: Dexketoprofen
Drug: Ibuprofen — third group: 400 mg Ibuprofen (İntrafen 400 mg vial-Gen-İstanbul) intravenous (IV) was given 70 patients, which determined to be applied as a group.
  Other Names: İntrafen
  Arms: Ibuprofen

SUMMARY:
* Currently, paracetamol and nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of patients with Acute Migraine Attack Headache
* The objective of the study is compare the efficacy of intravenous dexketoprofen,ibuprofen with paracetamol in the treatment of acute Migraine Attack Headache

DETAILED DESCRIPTION:
* This is the randomized double blinded clinical trial to compare the efficacy of these three drugs in this clinical setting.
* A randomized clinical trial was conducted in the Emergency Department (ED) of Pamukkale University Medical Faculty Hospital
* Study personnel (emergency physicians and nurses) were trained before the study.
* When intravenous drugs (Paracetamol, Dexketoprofen and ibuprofen) was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial Acute Migraine Attack Headache severity ratings with visual analog scale (VAS) were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of three groups:

First Group: 1000 mg of paracetamol ( perfalgan 10mg/ml solutionBristol- Myers Squibb_UK) intravenous (IV) was given 70 patients, Second Group: dexketoprofen 50 mg ( arveles ampoule -Ufsa- Istanbul) intravenous (IV) was given 70 patients, third group: 400 mg İbuprofen (İntrafen 400 mg vial-Gen-İstanbul) intravenous (IV) was given 70 patients, which determined to be applied as a group.

In addition, intravenous metoclopramide was added to the threatment of patients with acute migraine attack headache.

Drug packs prepared in 150 ml serum physiology were numbered by an independent nurse, who not involved in the study.

* Drugs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the paracetamol,dexketoprofen,ibuprofen medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered intravenously.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the acute migraine attack headache scores.
* Patients in three groups received three types of medication in a similar manner, thus ensuring double blind.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for inclusion if they were aged 18 years or older, 65 years or younger
* Isolated Migraine Attack Headache
* Patients who agree to work and receive the approval
* VAS (visual analog scale) score>5.

Exclusion Criteria:

* Patients with severe liver, kidney,pulmonary and cardiac heartfailure
* To be Pregnancy and breast-feeding
* Have received analgesics in the last 6hours
* Patients of childbearing age who are not using a birth control method.
* Patients with neurological deficits
* Patients with cardiac chest pain
* Patients with chronic pain
* Patients with pre-existing ibuprofen, dexketoprofen and paracetamol-induced gastrointestinal bleeding and perforation
* Patients with reflected pain
* Patients with neoplastic pain
* Patients with an allergy trait (ibuprofen, paracetamol and dexketoprofen)
* Illiterates and patients with vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
Decrement of the pain on VAS | Baseline and 60 minutes
  Comparison of the reduction of Migraine Attack Headache VAS (visual analog scale) score between the three groups. - (First group Paracetamol, Second Dexketoprofen and Third Ibuprofen )

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Turkcuer, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No